CLINICAL TRIAL: NCT01539057
Title: A Multicenter, Placebo Controlled Study to Evaluate the Efficacy of the Administration of Fibrinogen on Blood Product Requirements in Liver Transplantation
Brief Title: The Efficacy of the Administration of Fibrinogen in Liver Transplantation
Acronym: FibstudLT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Principal Investigator, Antoni Sabate, Head of Anesthesiology, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Promotor Code 1553-H-459; 2010-024584-41 (EudraCT Number)
Record Dates: First submitted 2012-02-02; First posted 2012-02-27 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Intraoperative Bleeding
Keywords: Liver; Surgery; hemostasis; coagulation; Fibrinogen
MeSH Terms: conditions — Blood Loss, Surgical; Thrombosis | interventions — Fibrinogen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Fibrinogen (Experimental): Fibrinogen will be administered until an expected plasmatic value of 2.9 g / L is achieved.
  Interventions: Drug: Fibrinogen
- Saline Serum (Placebo Comparator): the same dose in volume of saline dilution will be administered. The potential dose of fibrinogen required to obtain a final plasmatic reading of 2.9 g / L. will be computed. A serum will contain the corresponding ml of saline dilution
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Fibrinogen — The dose of fibrinogen should be calculated at 1 g of fibrinogen in order to obtain an increase in plasma fibrinogen value of 0.29 g / L to reach a final value of 2.9 g / L.
  Fibrinogen ampoules powder prepared with water dilution and located in a serum at a concentration of 2g/100 ml, which will be administered by intravenous infusion for 10 minutes.
  Administration before surgery starts
  Other Names: Haemocomplettan; RiaSTAP
  Arms: Intravenous Fibrinogen
Drug: Saline — the same dose in volume of water dilution will be administered. The potential dose of fibrinogen required to obtain a final plasmatic reading of 2.9 g / L. will be computed. A serum will contain the corresponding ml of water dilution. Administered before surgery starts
  Other Names: physiologic serum
  Arms: Saline Serum

SUMMARY:
Objective:

* To evaluate the efficacy of preoperative administration of fibrinogen in liver transplantation by maintaining a preoperative plasma level equal to 2.9 g / L compared with placebo, reflecting a reduction in the number of RBC units transfused during the procedure.
* To determine the influence of fibrinogen administration on mortality and survival of liver graft evaluated one year after the procedure.
* To determine the safety of fibrinogen administration recording thrombotic complications evaluated during hospitalization or at least 30 days postoperatively.

DETAILED DESCRIPTION:
Methods: A multicenter, randomized, double-blind, placebo-controlled study. One hundred thirty two patients (132) will randomly be assigned to:

Treatment group, Fibrinogen administration; doses of fibrinogen: 1 g for an increase in the plasmatic value of fibrinogen of 0.29 g / L to obtain a value of 2.9 g / L.

Placebo group, to whom the same dose volume of saline will be administered.

Determinations of haematocrit, electrolytes and kidney function tests and coagulation and haemostasis and thrombelastography test are made at all stages of the proceeding. A standard protocol for intraoperative management will be applied. Blood loss, administration of blood products, fluid therapy, presence of reperfusion syndrome, operative complications and mortality and survival will be registered. Patients will be followed for one year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for liver transplantation
* Patients with a value of pre-transplant plasma fibrinogen less than 2.9 g / L.

Exclusion Criteria:

* Patients with a value of fibrinogen in the 24 hours prior to the intervention than 2.9 g / L.
* Known history of thromboembolic events in 30 days
* Known or suspected pregnancy
* Previous randomization in this trial
* Known or suspected allergy to trial products or related products
* Known presence of congenital bleeding disorder. Patients treated with aspirin, warfarin
* The following indications for transplantation: familial polyneuropathy, acute liver failure, biliary cirrhosis and sclerosing cholangitis, Budd-Chiari syndrome
* Heart beating donors and living donor
* Patient reluctant to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients requiring transfusion of packed red blood cells during the procedure | intraoperative
  record of number of red blood cell packeds transfused during the surgical procedure

SECONDARY OUTCOMES:
Percentage of patients requiring blood products other than red cell concentrates | intraoperative
  * Number of packed red cells transfused during surgery
  * Number of units of fresh frozen plasma transfused during surgery
  * Number of platelet units transfused during surgery
  * Grams of fibrinogen administered during surgery
Operative outcome | 4 weeks
  * Operative mortality
  * Liver graft survival
  * Thrombotic complications of all types and causes
liver transplantation outcome | 1 year
  Follow-up of graft survival and patient mortality one year after liver transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Sabate, MD, Study Director — Hospital Universitari Bellvitge.IDIBELL
Locations (4):
- Spain (4):
  - Hospital Universitari de Bellvitge, Barcelona, Barcelona
  - Hospital Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Virgen del Rocio, Seville, Sevilla
  - Hospital de Cruces, Bilbao, Vizcaya

REFERENCES:
- [Derived] Perez L, Sabate A, Gutierrez R, Caballero M, Pujol R, Llaurado S, Penafiel J, Hereu P, Blasi A. Risk factors associated with blood transfusion in liver transplantation. Sci Rep. 2024 Aug 16;14(1):19022. doi: 10.1038/s41598-024-70078-2. PMID 39152310
- [Derived] Caballero M, Sabate A, Perez L, Vidal J, Reverter E, Gutierrez R, Crespo G, Penafiel J, Blasi A. Factors associated with mechanical ventilation longer than 24 h after liver transplantation in patients at risk for bleeding. BMC Anesthesiol. 2023 Nov 2;23(1):356. doi: 10.1186/s12871-023-02321-8. PMID 37919695
- [Derived] Blasi A, Sabate A, Beltran J, Costa M, Reyes R, Torres F. Correlation between plasma fibrinogen and FIBTEM thromboelastometry during liver transplantation: a comprehensive assessment. Vox Sang. 2017 Nov;112(8):788-795. doi: 10.1111/vox.12598. Epub 2017 Oct 8. PMID 28990201
- [Derived] Sabate A, Gutierrez R, Beltran J, Mellado P, Blasi A, Acosta F, Costa M, Reyes R, Torres F. Impact of Preemptive Fibrinogen Concentrate on Transfusion Requirements in Liver Transplantation: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial. Am J Transplant. 2016 Aug;16(8):2421-9. doi: 10.1111/ajt.13752. Epub 2016 Mar 17. PMID 26880105